CLINICAL TRIAL: NCT01107600
Title: Study on Immediate Loading of Immediately Placed Single Implants in Extraction Sockets With Nobel Active™ Implants and Bio-oss®.
Brief Title: Study on Immediate Loading of Immediately Placed Single Implants.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator and sponsor did not reach an agreement.
Sponsor: Hospital San Pietro Fatebenefratelli (Other)
Collaborators: Nobel Biocare (Industry); Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Marco Tallarico, Lecturer, Hospital San Pietro Fatebenefratelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSPFBF-NB-02
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Dental Implants
Keywords: Dental Implants, Single-Tooth; Bone Regeneration; Dental Restoration; Socket preservation

STUDY DESIGN:
Intervention Model Description: Immediate loading
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nobel Active® (Experimental): Immediate implant and socket preservation
  Interventions: Procedure: Immediate implant and socket preservation

INTERVENTIONS:
Procedure: Immediate implant and socket preservation — Implant placed in fresh extraction sockets as part of the same surgical procedure, and placed into occlusal loading within 48 h of implant placement. Guided bone regeneration with Biomaterial to preserve bone loss after tooth extraction.

SUMMARY:
The purpose of this study is to evaluate survival and success rates of dental implants placed with immediate loading protocol in extraction sockets. All patients were monitored for 1 year after implants placement.

DETAILED DESCRIPTION:
The international literature supported the potential advantages offered by this approach, but indicated a higher risk when compared with immediate loading in healed ridges.

The hypothesis to demonstrate is an high success and survival rates of Nobel Active™ implants used in combination with Bio-Oss® material.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Single-tooth implant restorations in the aesthetic zone

Exclusion Criteria:

* Medical risk patient
* Smoking

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06 (Estimated); Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Implant stability quote (ISQ) measurements. | 8 weeks
  Measured by Ostell® Mentor Device.

SECONDARY OUTCOMES:
Aesthetic Results and Patient Satisfaction | 1 year
  Bone crest level changes measured by standardized intraoral radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Gargari, Professor, Study Director — San Pietro Hospital, FBF, Roma
Locations (2):
- Italy (2):
  - Marco Tallarico, Rome
  - Odontoiatric center San Pietro Hospital, FBF, Rome

REFERENCES:
- [Background] Atieh MA, Payne AG, Duncan WJ, Cullinan MP. Immediate restoration/loading of immediately placed single implants: is it an effective bimodal approach? Clin Oral Implants Res. 2009 Jul;20(7):645-59. doi: 10.1111/j.1600-0501.2009.01725.x. PMID 19515058